CLINICAL TRIAL: NCT05369390
Title: Safety, Tolerability and Pharmacokinetics of NNC0487-0111 in Participants With Overweight or Obesity
Brief Title: A Research Study on How NNC0487-0111 Works in People With Overweight or Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9487-4830; U1111-1270-0852 (Other: World Health Organization (WHO))
Record Dates: First submitted 2022-05-04; First posted 2022-05-11 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Obesity
Keywords: overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: Single ascending dose (SAD) (Experimental): Participants will receive a single dose of any of the six different dose levels (1, 3, 6, 12, 25 and 50 milligrams (mg)) of NNC0487-0111 A or matching placebo in a sequential manner with the dose increasing between cohorts.
  Interventions: Drug: NNC0487-0111 A; Other: Placebo A (NNC0487-0111 A)
- Part B: Multiple ascending dose (MAD) (Experimental): Participants will receive NNC0487-0111 once daily for 10 days at any of the five different dose levels (3, 6, 12, 25 and 50 milligrams (mg)) of NNC0487-0111 A or matching placebo in a sequential manner with the dose increasing between cohorts.
  Interventions: Drug: NNC0487-0111 A; Other: Placebo A (NNC0487-0111 A)
- Part C (Experimental): Participants will receive NNC0487-0111 A or matching placebo once-daily for 12 weeks: 3 or 6 mg for weeks 1-2, 6 or 12 mg for weeks 3-4, 12 or 25 mg for weeks 5-6, 25 or 50 mg for weeks 7-8, 25 or 50 mg for weeks 9-10 and 50 or 2*50 mg for weeks 11-12.
  Interventions: Drug: NNC0487-0111 A; Other: Placebo A (NNC0487-0111 A)
- Part D (Experimental): Participants will receive NNC0487-0111 B or matching placebo once-daily for 12 weeks: 3 or 6 mg for weeks 1-2, 6 or 12 mg for weeks 3-4, 12 or 25 mg for weeks 5-6, 25 or 50 mg for weeks 7-8, 25 or 50 mg for weeks 9-10 and 50 or 2*50 mg for weeks 11-12.
  Interventions: Drug: NNC0487-0111 B; Other: Placebo B (NNC0487-0111 B)

INTERVENTIONS:
Drug: NNC0487-0111 A — Participants will receive NNC0487-0111 A tablet once daily.
  Arms: Part A: Single ascending dose (SAD); Part B: Multiple ascending dose (MAD); Part C
Drug: NNC0487-0111 B — Participants will receive NNC0487-0111 B tablet once daily.
  Arms: Part D
Other: Placebo B (NNC0487-0111 B) — Participants will receive placebo matched to NNC0487-0111 B tablet once daily.
  Arms: Part D
Other: Placebo A (NNC0487-0111 A) — Participants will receive placebo matched to NNC0487-0111 A tablet once daily.
  Arms: Part A: Single ascending dose (SAD); Part B: Multiple ascending dose (MAD); Part C

SUMMARY:
NNC0487-0111 is a new medicine similar to 2 hormones that are produced in human body: amylin and glucagon-like peptide-1 (GLP-1). Both hormones work like body's own hormones and help the body to feel full. This study tests if the study medicine is safe and to find out how the medicine works in humans. This study also look at how the study medicine affects body weight and how to improve the treatment of people with overweight, obesity or related diseases.

This study will have 4 parts: Part A, B, C and D. Part A: This is planned to consist of five groups, one additional group may be added. Each group will include 8 participants, with 6 participants being randomised to receive a single dose of NNC0487-0111 A and 2 participants randomised to receive placebo. The dosing within each group will be sequential, i.e., 2 sentinel participants (1 on active and 1 on placebo).

Part B: This is planned to consist of three groups, one additional group may be added. Each group will include 12 participants, with 9 participants being randomised to receive NNC0487-0111 A and 3 participants randomised to receive placebo once daily for 10 days. The dosing within each group will be sequential. For the first group, 4 sentinel participants (3 on active and 1 on placebo) will be dosed followed by a safety observation period of 7 days (168 hours), before dosing of the remaining participants in the group will be initiated. For the remaining groups, 4 sentinel participants (3 on active and 1 on placebo) will be dosed followed by a safety observation period of at least 36 hours before dosing of the remaining participants in the group will be initiated.

Part C and D are matching regarding planned visits and procedures, but the study interventions in Part D (NNC0487-0111 B) differ from Part A, B and C (NNC0487-0111 A). Each part is planned to consist of one group, although one additional group may be added. Each group will include 20 participants, with 16 participants being randomised to receive active treatment and 4 participants randomised to receive placebo once-daily for 12 weeks. The dosing will be sequential, i.e., 4 sentinel participants (3 on active and 1 on placebo) will be dosed followed by a safety observation period of at least 36 hours before dosing of the remaining participants in the cohort will be initiated. The remaining participants will be dosed in smaller groups of 8 participants separated by a safety observation period of at least 36 hours.

A safety evaluation will be made between dosing of participants within a group and before moving on to a higher dose.

ELIGIBILITY:
Inclusion Criteria:

Part A and B:

* Male or female aged 18-55 years (both inclusive) at time of signing informed consent
* Body mass index (BMI) of 25.0 to 34.9 kilogram per square meter (kg/m^2) (both inclusive) at screening
* Considered eligible based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Part C and D:

* Male or female aged 18-55 years (both inclusive) at time of signing informed consent
* Body mass index (BMI) of 27.0 to 39.9 kg/m^2 (both inclusive) at screening
* Considered eligible based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

Part A and B:

* Any disorder, which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol
* HbA1c greater than or equal to 6.5 % (48 millimoles per mole (mmol/mol)) at screening
* Any laboratory safety parameters at screening outside the below laboratory ranges, see designated reference range documents for specific values
* Vitamin D (25-hydroxycholecalciferol) less than 20 Nanograms per milliliter (ng/mL) (50 nano molar (NM)) at screening
* Parathyroid hormone (PTH) outside normal range at screening
* Total calcium outside normal range at screening
* Amylase greater than or equal to 2 times upper limit of normal at screening
* Lipase greater than or equal to 2 times upper limit of normal at screening

Part C and D:

* Any disorder, which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol
* HbA1c greater than or equal to 6.5 % (48 mmol/mol) at screening
* Any laboratory safety parameters at screening outside the below laboratory ranges, see designated reference range documents for specific values:
* Vitamin D (25-hydroxycholecalciferol) less than 20 ng/mL (50 nM) at screening
* Parathyroid hormone (PTH) outside normal range at screening
* Total calcium outside normal range at screening
* Amylase greater than or equal to 2 times upper limit of normal at screening
* Lipase greater than or equal to 2 times upper limit of normal at screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-01-09 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAE) | Part A: From pre-dose on Day 1 to 22 days; Part B: From pre-dose on Day 1 to 31 days; Part C and D: From pre-dose on Day 1 to 105 days
  Number of events

SECONDARY OUTCOMES:
Part A: AUC0-∞,SD; the area under the NNC0487-0111 plasma concentration-time curve from time 0 to infinity after a single dose | From pre-dose on Day 1 until completion of the end of study visit (Day 22)
  Hours*Nanomoles per liter (h*nmol/L)
Part A: Cmax,SD; the maximum plasma concentration of NNC0487- 0111 after a single dose | From pre-dose on Day 1 until completion of the end of study visit (Day 22)
  Nanomoles per liter (nmol/L)
Part B: AUC0-24h,MD; the area under the NNC0487-011 plasma concentration-time curve from time 0 to 24 hours after last multiple dose | From pre-dose on Day 10 until Day 11 (24 hours post-dose)
  h*nmol/L
Part B: Cmax,MD; the maximum plasma concentration of NNC0487- 0111 after last multiple dose | From pre-dose on Day 10 until Day 22
  nmol/L
Part C and D: AUC0-24h,MD; the area under the NNC0487-011 plasma concentration-time curve from time 0 to 24 hours after last multiple dose | From pre-dose on Day 84 until Day 85 (24 hours post-dose)
  h*nmol/L
Part C and D: Cmax,MD; the maximum plasma concentration of NNC0487- 0111 after last multiple dose | From pre-dose on Day 84 until completion of the end of study visit (Day 105)
  nmol/L

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - ICON Early Phase Services, LLC, San Antonio, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Gasiorek A, Heydorn A, Gabery S, Hjerpsted JB, Kirkeby K, Kruse T, Petersen SB, Toubro S, Vegge A, Key C. Safety, tolerability, pharmacokinetics, and pharmacodynamics of the first-in-class GLP-1 and amylin receptor agonist, amycretin: a first-in-human, phase 1, double-blind, randomised, placebo-controlled trial. Lancet. 2025 Jul 12;406(10499):135-148. doi: 10.1016/S0140-6736(25)01176-6. Epub 2025 Jun 20. PMID 40550229